

Statistical Analysis Plan for Masimo Study titled "Calibration and Validation of Masimo's O3 Regional Oximetry Device in Neonates, Infants and Children Undergoing Cardiac Catherization"

**Protocol Date:** 9 MAY 2018

NCT Number: NCT03123354

Statistical Analysis Plan for Masimo Study titled "Calibration and Validation of Masimo's O3 Regional Oximetry Device in Neonates, Infants and Children Undergoing Cardiac Catherization"

## **Data Analysis**

We compute error statistics, including mean bias, precision, standard deviation of bias, and absolute root-mean-squared-error accuracy  $A_{rms}$ , accounting for within-subject correlations.

## **Applicable Analysis Methods**

Measurement error or bias for the kth sample e(k) is defined as

$$e(k) = rSO_2(k) - SavO_2(k)$$
.

Mean bias over N data points is defined as

$$\mu = \frac{1}{N} \sum_{k=1}^{N} e(k)$$

The A<sub>rms</sub> can be calculated as

$$A_{rms} \approx \sqrt{\mu^2 + s^2}$$

where s is the estimated standard deviation of bias, accounting for within-subject correlation, which is calculated using the Bland and Altman method for repeated measures. The 95% confidence interval of mean bias was calculated as  $(\mu - 2s/\sqrt{N})$ .